CLINICAL TRIAL: NCT04655547
Title: Impact on Energy Intake by Implementing Recommended Food Texture Through Dietary Guidance at the Department of Swallowing and Eating Disorders; a Randomized Clinical Trial
Brief Title: Impact on Energy Intake by Implementing Recommended Food Texture Through Dietary Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS19953
Record Dates: First submitted 2020-11-24; First posted 2020-12-07 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-08

CONDITIONS: Energy Intake; Activities of Daily Living; Quality of Life; Protein Intake; Fluid Balance; Lean Body Mass; Fat Mass; Weight
Keywords: Dysphagia; Dietary Guidance; Energy- and Protein intake; Food Texture; Activities of Daily Living and Quality of Life
MeSH Terms: conditions — Body Weight; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to control or intervention group, stratified on their FEDSS-score.
  The study will include 34 participants - 17 in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The participants will follow the usual offered course on the outpatient clinic of Hammel Neurocenter. They wil anticipate in data collection three times in line with the intervention group.
- Intervention (Experimental): The participants will receive dietary guidance from an dietician, with focus on energy intake and food texture. This guidance will include two sessions on site and three phone meetings. The last on site meeting, will be concluding.
  Interventions: Other: Dietary guidance

INTERVENTIONS:
Other: Dietary guidance — Dietary guidance with focus on texture and energy intake, preformed by certified dietitians.
  Arms: Intervention

SUMMARY:
An intervention study on the effect of dietary guidance with focus on implementing recommended food texture, at the department of Eating and Swallowing difficulties, Region Midtjylland, Denmark.

Energy- and protein intake, Weightloss, Bodymass composition, Fluid balance and Activities of Daily Living (ADL), will be measured by Bioimpedance spectroscopy, interviews and a questionnaire.

DETAILED DESCRIPTION:
It is know that people with eating- and swallowing difficulties(known as dysphagia), is prone to weightloss due to insufficient energy- and protein intake, and a reduction in ADL.

ADL will in this project have its focus on the eating situation.

The projects research questions are:

* Will dietary guidance with texture implementation increase energy intake in patients being examined on an outpatient basis for dysphagia, based on the Fiberoptic Endoscopic Evaluation of Swallowing (FEES) recommendation?
* Can a dietetic guidance with texture implementation increase quality of life and ADL in patients with dysphagia?

Recruitment and data collection will take place at Hammel Neurocenter, DK.

Each patient will be included for eight weeks, after their first FEES examination. The participants will be randomized to control or intervention, and strata into three groups based on Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) 1, 2-3 and 4.

Within the eight weeks, participants have to show up three times to measurements, interviews and questionnaire, in addition to this, the intervention groups will have three follow-up phone meetings.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Newly refered patients to FEES examination
* Score 1-4 on FEDSS-scale
* Consumes 50% energy or more orally
* Consumes less energy than calculated energy need (Harris-Benedict)
* Individuals of full legal capacity
* Individuals above 18 of years
* That the patient is capable of executing examinations

Exclusion Criteria:

* Individuals with known eating disorders
* Ineligible individuals
* Individual in need of translator
* Individuals participating in another trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in energy intake, from baseline. | Eight weeks
  Change in energy intake, measured from baseline. Measured in kilojoule by a standardized interview with examples of pictures to determine serving size.

SECONDARY OUTCOMES:
Changes in Dysphagia Handicap Index (DHI) total and section (E and F) score. | Eight weeks
  DHI is a questionnaire with 25 questions, divided into three sections. possible scores are minimum 25 and maximum 125. The higher the score, the worse dysphagia status.
  Measured in points, changes from baseline.
In how many questions in the DHI, does the intervention group change the score in relation to the control group, and with how much. | Eight weeks
  Measured in points, changes from baseline.
Body Weight. | Eight weeks
  Measured in kilograms, by bioimpedance spectroscopy, changes from baseline.
Lean Body Mass. | Eight weeks
  Measured in kilograms, by bioimpedance spectroscopy, changes from baseline.
Fat Mass. | Eight weeks
  Measured in kilograms, by bioimpedance spectroscopy, changes from baseline.
Fluid Balance. | Eight weeks
  Measured in kilograms, by bioimpedance spectroscopy, changes from baseline.
Changes in protein intake. | Eight weeks
  Measured in gram, by a standardized interview with examples of pictures to determine serving size, from baseline.
Compliance of recommended changes. | Eight weeks
  Measured by score through interview. Minimum score 1 and maximum score 5. The greater the score, the better compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Fabricius, Ph.d., Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Central Jutland, Denmark